CLINICAL TRIAL: NCT04125693
Title: A Roll-over Study to Provide Continued Treatment With Rogaratinib in Participants Who Were Enrolled in Rogaratinib Studies
Brief Title: Roll-over Study to Continue Treatment With the Investigational Drug Rogaratinib and to Further Test Its Safety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20252; 2019-000808-15 (EudraCT Number)
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: Fibroblast growth factor receptors (FGFR) Inhibitor; FGFR 1-4; Non-small-cell lung cancer; Small-cell lung cancer; Urothelial carcinoma; Adenoidcystic carcinoma; Head cancer; Neck cancer; Breast cancer
MeSH Terms: conditions — Neoplasms; Acrocephalosyndactylia; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Transitional Cell; Head and Neck Neoplasms; Breast Neoplasms | interventions — Rogaratinib; Drug Combinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients (Experimental): Patients from completed Bayer clinical trials, who received rogaratinib as monotherapy or combination therapy for the treatment of cancer.
  Interventions: Drug: Rogaratinib (BAY1163877); Drug: Combination drug

INTERVENTIONS:
Drug: Rogaratinib (BAY1163877) — Participants will be treated with investigational drug following the treatment schedule and dosing instructions from the feeder-study protocol.
  Other Names: FGFR 1-4 inhibitor
Drug: Combination drug — Any other drug specified in the protocol of the completed Bayer clinical trials that is used in combination with rogaratinib. Not all patients receive combination therapy.

SUMMARY:
The purpose of this study is to enable patients, who are currently receiving rogaratinib in a Bayer-sponsored clinical trial (incl. NCT01976741), to continue treatment after their respective study has been closed. Another aim is to learn if rogaratinib is safe and how it affects the body.

Rogaratinib is an investigational drug that may treat different types of cancer, incl. non-small-cell lung cancer, small-cell lung cancer, urothelial carcinoma, head, neck and breast cancer. The drug may stop the growth of cancer cells by targeting different cell proteins called fibroblast growth factor receptors (FGFR) that are needed for the survival of the cancer cells.

DETAILED DESCRIPTION:
The primary objectives of the study are the continuation of rogaratinib treatment (as monotherapy or combination therapy) for patients after closure of their feeder studies and the further assessment of the safety of the drug.

The secondary objective is to investigate the tolerability of rogaratinib.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in any Bayer-sponsored rogaratinib feeder study at the time of study closure, who are currently receiving rogaratinib (monotherapy or combination therapy) and are experiencing clinical benefit from treatment, determined by the treating physician.
* Participants who meet criteria to initiate a subsequent cycle of therapy, as determined by the guidelines of the feeder study protocol.
* Any ongoing adverse events that required temporary treatment interruption must be resolved to baseline grade or assessed as stable and not requiring further treatment interruption.
* Women of childbearing potential and men with reproductive potential must be willing to continue practicing acceptable methods of birth control during the study treatment and until 6 months after stopping study treatment.

Exclusion Criteria:

* Ineligibility, for medical reasons, to start the next treatment cycle in the respective feeder study.
* Patients with a beta-human chorionic gonadotropin (hCG) test consistent with pregnancy.
* Participants are using one or more of the prohibited medications listed in the respective feeder study protocol
* Negative benefit / risk ratio as determined by the investigator
* Positive pregnancy test for on-treatment participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 55 months
Incidence of treatment-emergent serious adverse events (TESAEs) | Up to 55 months
Incidence of drug-related TEAEs | Up to 55 months
Incidence of drug-related TESAEs | Up to 55 months

SECONDARY OUTCOMES:
Frequency of dose modifications | Up to 55 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.